CLINICAL TRIAL: NCT04340817
Title: Fatty Liver Disease in Nordic Countries (FLINC): a Prospective Cohort Study
Brief Title: Fatty Liver Disease in Nordic Countries
Acronym: FLINC
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Lise Gluud, Professor, Copenhagen University Hospital, Hvidovre
Other Study IDs: Flinc07042020
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Genome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, buffy coat, liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Proteomics — Mass-spectometry proteomics
Diagnostic Test: Transcriptomics — Next generation sequencing
Genetic: Genomics — Targeted genetics

SUMMARY:
A prospective cohort study, which aims to systematically evaluate biomarkers and potential targets in NAFLD and NASH.

ELIGIBILITY:
Inclusion Criteria:

* Non-alcoholic fatty liver disease and
* Healthy volunteers

Exclusion Criteria:

* Other liver diseases than non-alcoholic fatty liver disease
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to include patients with suspected or verified non-alcoholic fatty liver disease
Sampling Method: Non-Probability Sample
Enrollment: 634 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Fibrosis | 5 years
  Number of participants with fibrosis proression

CONTACTS AND LOCATIONS:
Overall Officials: Lise L Gluud, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Gastrounit, Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided